CLINICAL TRIAL: NCT06783374
Title: Effect of a Peripheral and Central Neuromodulation Protocol Combined With the Application of Therapeutic Exercise in Patients Diagnosed With Urinary Incontinence. A Randomized Control Trial (RCT)
Brief Title: Effect of Neuromodulation and Therapeutic Exercise in Urinary Incontinence
Acronym: UCV/INCONTINEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCV/2024-2025/020; Ethical Commithe (Other: FundacionUCV)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-12

CONDITIONS: Urge Urinary Incontinence; Overactive Bladder (OAB)
Keywords: Menopause; exercise; Neuromodulation; Posterior tibial nerve
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive; Motor Activity | interventions — Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The groups will be arranged randomly, and the masking technique to be employed will be a double-blind procedure. The subjects will be randomly selected utilizing the EPIDAT 3.1 program. Both the participants and the investigator responsible for data collection remained unaware of the assigned intervention and the results obtained, respectively, until the study's conclusion. An independent researcher, employing an Excel formula, generated a table of random numbers to blind data collectors and outcome adjudicators, thereby ensuring unbiased outcome ascertainment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exercise + neuromodulation (Experimental): The Intervention group will initially undergo posterior tibial nerve neuromodulation following a standardized protocol: 30 minutes per session, 2 sessions per week for 3 months. Sessions will have a duration of 60 minutes and will be structured into three distinct blocks. In the initial two treatment blocks, exercises will emphasize CORE stabilization and general strength training with forced exhalation to ensure appropriate activation of the transverse abdominal muscle, with the objective of preventing adverse effects associated with increased intra-abdominal pressure. The third work block will focus on addressing anticipatory postural adjustment control, given its established relationship with the pelvic floor muscles. This technique will be actively implemented in conjunction with the Proprioceptive Postural Reeducation Method (5P® LOGSURF).
  Interventions: Procedure: Neuromodulation; Procedure: Exercise
- Exercise+ ShamNeuromodulation (Sham Comparator): For the SHAM group, a non-penetrating needle with a retractable handle will be utilized, which is commonly employed in experimental research with Streitberger and Kleinhenz placebo needles. This method creates the appearance of insertion without penetrating the skin and allows the needles to remain in situ for the duration of the intervention. The SHAM group participants will adhere to the exercise protocol in the same manner as the intervention group.
  Interventions: Procedure: Exercise; Procedure: Sham Neuromodulation
- Control Group (Active Comparator): Conventional Physiotherapy. The control group engages in specific pelvic floor exercises, which are less complex in terms of neuromuscular processing (focusing on fundamental spinal stimuli), in contrast to the more comprehensive and intricate tasks of the intervention group. Additionally, manual therapy techniques are employed to inhibit trigger points in the musculature and ligamentous structures of the pelvic cavity, as well as intracavitary techniques aimed at alleviating mechanical pain.
  Interventions: Procedure: Exercise control group

INTERVENTIONS:
Procedure: Neuromodulation — A protocol of posterior tibial nerve electrostimulation will be implemented, inducing retrograde electrostimulation through the pelvic nerves, which are connected to the spinal cord via the sacral plexus at segments S2 and S3. It is recommended to conduct an average of 10 sessions to evaluate the efficacy of the treatment, within a range of 6 to 16 sessions, each lasting 30 minutes, completing a treatment period of 3 months.
  Arms: Exercise + neuromodulation
Procedure: Exercise — Participants will engage in a 60-minute exercise session, divided into two blocks: Block 1 will comprise 10 to 12 repetitions per set, aiming to achieve a perceived exertion level of 7 to 10 on the rating of perceived exertion (RPE). Block 2 will utilize the 5P® LOGSURF Method, termed Proprioceptive Perineal Postural Reeducation, which employs unstable positions to promote postural adjustment and continuous balance. This approach facilitates the activation of the abdominopelvic muscles, enhancing control and strengthening of the pelvic-perineal region.
  Arms: Exercise + neuromodulation; Exercise+ ShamNeuromodulation
Procedure: Exercise control group — Exercise The control group engages in specific pelvic floor exercises, which are less complex in terms of neuromuscular processing, such as Kegel's exercise. The protocol for these exercises is standardized and conducted individually, comprising 8 to 12 sessions of 20-40 minutes each, performed twice weekly.
  Arms: Control Group
Procedure: Sham Neuromodulation — A needle with a retractable handle will be used, commonly employed in experimental research with Streitberger and Kleinhenz placebo needles. This creates the appearance of insertion without penetrating the skin and allows the needles to remain in place for the duration of the intervention.
  Arms: Exercise+ ShamNeuromodulation

SUMMARY:
Urge urinary incontinence (UUI) is a component of the condition known as overactive bladder, a severe and debilitating chronic disorder affecting healthcare systems worldwide. The efficacy of therapeutic exercise and neuromodulation in the treatment of UUI is evaluated, and these techniques are combined.

DETAILED DESCRIPTION:
Urge urinary incontinence (UUI) is a component of the condition known as overactive bladder, a severe and debilitating chronic disorder that affects the neurophysiology of micturition and bladder functionality, particularly in processes associated with menopause, leading to a deterioration in quality of life. Various therapeutic approaches are employed to treat overactive bladder. Among the most frequently implemented interventions are sacral or tibial nerve neurostimulation. This intervention targets the pathophysiological substrate by modulating the somatic afferent activity of the bladder and interfering with the activity of fibers responsible for pain modulation and neuromuscular system functionality. In essence, the described approach focuses on reducing peripheral input. Based on the aforementioned information, it was hypothesized that training through a pelvic floor strength protocol, performed adjunctively with peripheral neuromodulation prior to its implementation, may provide the ability to inhibit detrusor contractions via involuntary contractions of the perineal musculature.

ELIGIBILITY:
Inclusion Criteria:

* Present with a diagnosis of urinary incontinence or overactive bladder
* Women of menopausal age (>45 years)
* ≥3 months of duration
* Fulfill the established criteria for patient selection for neuromodulation treatment (urge urinary incontinence)
* Speak native Spanish or English

Exclusion Criteria:

* Prior or scheduled surgical procedures in the lumbar or abdominal region
* Presence of fractures or severe pathological conditions
* Current pregnancy or potential for pregnancy during the study period
* Neurological or psychiatric disorders
* Presence of stress urinary incontinence
* Female subjects with autoimmune diseases or malignancies
* Belonephobia
* Subjects who have undergone previous neuromodulation

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
The Overactive Bladder Questionnaire-Short Form | At baseline, Post1month, Post3months, Post6months
  The Overactive Bladder Questionnaire-Short Form (OAB-q SF) is a concise, self-administered patient-reported outcomes instrument comprising two scales that assess symptom bother and health-related quality of life (HR-QOL) in patients with OAB. This self-administered, disease-specific questionnaire evaluates symptomatic discomfort (6 items) and health-related quality of life (HRQoL, 13 items) using a 6-point Likert scale. Scores are transformed to a 0-100 scale, where higher symptom scores indicate greater severity, and higher HRQoL scores reflect better quality of life

SECONDARY OUTCOMES:
Mapping of Incontinence Quality of Life (I-QOL) | at baseline, Post1month, Post3months, Post6months
  Mapping of Incontinence Quality of Life (I-QOL) is a widely utilized self-reported health-related quality of life instrument for individuals with urinary incontinence (UI). It comprises 22 items, each employing a 5-point ordinal response scale where 1 = extremely, 2 = quite a lot, 3 = moderately, 4 = a little, and 5 = not at all.
Bladder Diary | at baseline, Post1month, Post3months, Post6months
  Bladder Diary is a non-invasive assessment tool that provides insights into bladder function. It is utilized to measure the frequency and severity of urinary dysfunction symptoms, such as overactive bladder.
Urinary Incontinence Short Form (ICIQ-UI-SF) | at baseline, Post1month, Post3months, Post6months
  Urinary Incontinence Short Form (ICIQ-UI-SF) comprises three components that assess subjective frequency, subjective severity, and quality of life through a self-administered questionnaire. Questions 3 to 5 are scored items, with responses totaled to achieve a minimum score of 0 and maximum of 21.
Electromyography (EMG) | at baseline, Post1month, Post3months, Post6months
  Electromyography (EMG) is a reliable, non-invasive method to assess pelvic floor muscle (PFM) tone, strength, endurance, and function. Electrical activity is recorded using a vaginal probe to monitor deep and superficial PFM layers. Measurements are obtained in supine and standing positions.
Oxford Scale | at baseline, Post1month, Post3months, Post6months
  Oxford Scale is a subjective classification system utilized to evaluate the strength and quality of pelvic floor muscle (PFM) contractions through intracavitary palpation with one or two fingers. The modified scale comprises 5 grades: 0 = no contraction; 1 = flickering muscle movements; 2 = weak contraction; 3 = increased pressure with slight muscle elevation; 4 = firm contraction with moderate elevation of the vaginal posterior wall; 5 = strong contraction with finger resistance against the abdominal wall.
Tampa Scale-11 (TSK-11) | at baseline, Post1month, Post3months, Post6months
  Tampa Scale-11 (TSK-11) is a validated instrument for assessing kinesiophobia, or fear of movement, in individuals with chronic pain. It identifies fear-avoidance beliefs with scores ranging from 11 to 44, where higher scores indicate greater fear of reinjury. The TSK-11 demonstrates reliability (α = 0.84) and is widely employed in musculoskeletal pain populations.
Pain Catastrophizing Scale (PCS) | at baseline, Post1month, Post3months, Post6months
  Pain Catastrophizing Scale (PCS) is a 13-item self-administered instrument assessing pain magnification, rumination, and helplessness. Scores range from 13 to 62, with higher scores indicating greater catastrophizing. The validated Spanish version exhibits high reliability (α = 0.95; test-retest r = 0.70-0.75).
Sport Injury Rehabilitation Adherence Scales (SIRAS) | at baseline, Post1month, Post3months, Post6months
  Sport Injury Rehabilitation Adherence Scales (SIRAS) evaluates patient adherence during rehabilitation sessions, as rated by healthcare professionals. It assesses the intensity with which patients complete exercises, their consistency in following instructions, and their receptiveness to program adjustments. The scale comprises three items scored to produce a total between 0 and 15, with higher scores indicating greater adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic Univerity of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuentes-Aparicio L, Arranz-Martin B, Navarro-Brazalez B, Bailon-Cerezo J, Sanchez-Sanchez B, Torres-Lacomba M. Postural Sensorimotor Control on Anorectal Pressures and Pelvic Floor Muscle Tone and Strength: Effects of a Single 5P(R) LOGSURF Session. A Cross-Sectional Preliminary Study. Int J Environ Res Public Health. 2021 Apr 2;18(7):3708. doi: 10.3390/ijerph18073708. PMID 33918217
- [Background] Sonmez R, Yildiz N, Alkan H. Efficacy of percutaneous and transcutaneous tibial nerve stimulation in women with idiopathic overactive bladder: A prospective randomised controlled trial. Ann Phys Rehabil Med. 2022 Jan;65(1):101486. doi: 10.1016/j.rehab.2021.101486. Epub 2021 Nov 11. PMID 33429090
- [Background] Arlandis S, Ruiz MA, Errando C, Villacampa F, Arumi D, Lizarraga I, Rejas J. Quality of life in patients with overactive bladder: validation and psychometric properties of the Spanish Overactive Bladder Questionnaire-short Form. Clin Drug Investig. 2012 Aug 1;32(8):523-32. doi: 10.2165/11633760-000000000-00000. PMID 22741748
- [Background] Fernandez-Cuadros ME, Martin-Martin LM, Albaladejo-Florin MJ, Perez-Moro OS, Alava-Rabasa S, Goizueta-San-Martin G. [Transcutaneous stimulation of the posterior tibial nerve modifies the sympathetic skin response and improves overactive bladder syndrome: Case series and possible diagnostic test]. Rehabilitacion (Madr). 2022 Oct-Dec;56(4):255-263. doi: 10.1016/j.rh.2021.04.005. Epub 2021 Sep 24. Spanish. PMID 34565565
- [Background] Bo K, Berghmans LC. Nonpharmacologic treatments for overactive bladder-pelvic floor exercises. Urology. 2000 May;55(5A Suppl):7-11; discussion 14-6. PMID 10767443
- [Background] Abrams P. Describing bladder storage function: overactive bladder syndrome and detrusor overactivity. Urology. 2003 Nov;62(5 Suppl 2):28-37; discussion 40-2. doi: 10.1016/j.urology.2003.09.050. PMID 14662404
- [Background] Carcelen-Fraile MDC, Aibar-Almazan A, Martinez-Amat A, Cruz-Diaz D, Diaz-Mohedo E, Redecillas-Peiro MT, Hita-Contreras F. Effects of Physical Exercise on Sexual Function and Quality of Sexual Life Related to Menopausal Symptoms in Peri- and Postmenopausal Women: A Systematic Review. Int J Environ Res Public Health. 2020 Apr 14;17(8):2680. doi: 10.3390/ijerph17082680. PMID 32295114
- [Derived] Leal-Garcia J, Blanco-Gimenez P, Jaenada-Carrillero E, Martinez-Soler M, Huertas-Ramirez B, Mahiques-Sanchis A, Vicente-Mampel J. Effect of a Peripheral Neuromodulation Protocol Combined with the Application of Therapeutic Exercise in Patients Diagnosed with Urinary Incontinence-A Study Protocol for a Randomized Controlled Trial. Healthcare (Basel). 2025 Jul 21;13(14):1759. doi: 10.3390/healthcare13141759. PMID 40724784